CLINICAL TRIAL: NCT06806527
Title: Validity and Reliability of the Six-minute Peg Board and Ring Test in Patients With Chronic Neck Pain
Brief Title: Validity and Reliability of the Six-minute Peg Board and Ring Test in Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Başak KAVALCI KOL, Principal Investigator, Kirsehir Ahi Evran Universitesi
Other Study IDs: AhiEvranU527
Record Dates: First submitted 2025-01-17; First posted 2025-02-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Chronic Neck Pain
Keywords: exercise capacity; six-minute peg board and ring test; chronic neck pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Neck Pain Group: Individuals between the ages of 18-65 who have had neck pain for at least 12 weeks and are being followed up at the Physical Therapy Polyclinic of the Physical Medicine and Rehabilitation Department of Kırşehir Ahi Evran University will be included in the study.

SUMMARY:
The purpose of this study was to evaluate the validity and reliability of six-minute peg board and ring test (6-PBRT) in individuals with chronic neck pain and to determine the applicability of the test for this patient population.

DETAILED DESCRIPTION:
Neck pain is the fourth leading cause of disability worldwide and is a significant public health problem. Chronic neck pain is defined as the presence of pain in the neck region of individuals for more than twelve weeks. Chronic neck pain is a disorder that negatively affects the individual's daily life activities and causes labor force and economic losses by causing functional limitations, loss of work and disability. It is important to evaluate the physical fitness components in detail in individuals with chronic neck pain. It has been stated that neck pain reduces upper extremity performance.

Different measurement methods have been used to evaluate the upper extremity functions of individuals. Standard measurement tools are needed to evaluate the upper extremity exercise capacity in patients with chronic neck pain. The 6-PBRT is a valid, reliable, useful, practical and easy-to-apply test that evaluates the endurance of the upper extremity without support in healthy individuals and those with chronic obstructive pulmonary disease. The validity and reliability of 6-PBRT, which is used to evaluate functional upper extremity exercise capacity in different diseases, has not been investigated in individuals with chronic neck pain. The aim of this study was to evaluate the validity and reliability of 6-PBRT in individuals with chronic neck pain and to determine the applicability of the test for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with neck pain that has lasted at least 3 months due to problems such as cervical strain or sprain, cervical disc lesions, cervical spondylosis, facet joint dysfunction and myofascial pain syndrome,
* Those between the ages of 18-65,
* Individuals who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Neck pain severity under 3 point during activity according to Visual Analog Scale
* Motor deficit in upper extremity neurological examination
* Undergone any surgery related to neck problem
* Presence of cervical radiculopathy
* Undergone any upper extremity surgery,
* Presence of rheumatic and/or neurological disease or any disease affecting the vestibular system
* Presence of carpal tunnel syndrome, rotator cuff syndrome, impingement syndrome, thoracic outlet syndrome, lateral and medial epicondylitis, hand osteoarthritis that will affect upper extremity and hand functions
* Individuals with cognitive dysfunction who will understand and apply the exercise test instructions will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are followed up in the Physical Therapy Polyclinic of the Physical Medicine and Rehabilitation Department of Kırşehir Ahi Evran University, between the ages of 18-65, who have neck pain for at least 12 weeks, and who meet the specified inclusion and exclusion criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Six-minute pegboard and ring test | First day and second day
  The six minute pegboard and ring test (6-PBRT) will be used to assess upper extremity exercise capacity. The test will be repeated twice on the first and second day evaluations. One week later, the second 6-PBRT test will be performed for reliability analysis.

SECONDARY OUTCOMES:
Maximal symptom-limited arm ergometer test | First day
  Maximal symptom-limited arm ergometer test will be performed to analyze the validity of the 6-PBRT. The test will be used as the criterion measure for the validity of the six minute peg board and ring test. For the test, the height of the ergometer will be adjusted to be at shoulder level and the test will be performed in a sitting position.
Hand-grip strength | Second day
  For validity the correlation between 6-PBRT and hand grip strength will be examined. Hand grip strength will be assessed using a hand dynamometer. Patients will sit in a 90° upright position with their knees, wrists in neutral, elbows at 90° and the dynamometer attached to the body will be grasped with all their strength. Measurements will be repeated 3 times on the right and left extremities with 10 seconds intervals and the highest value will be recorded. The percentage of expected values determined according to age and gender will be used in the interpretation of the measurements.
Disabilities of the arm, shoulder and hand (DASH) questionnaire | First day
  It will be used to evaluate the upper extremity functional status of patients. For validity, the correlation between 6-PBRT and functional status will be examined. Disabilities of the arm, shoulder and hand (DASH) questionnaire evaluates the functional status of the upper extremity subjectively according to the Likert scale. The scale consists of three parts. The questionnaire scores between 0 (no disability) and 100 (severe disability).
Evaluation of pain severity | First day
  The severity of the individuals' resting activity and night pain will be questioned with the Visual Analog Scale. The visual analog scale is a scale consisting of a horizontal line of 100 mm length, 0 mm meaning no pain and 100 mm meaning unbearable pain. Individuals will be asked to place a mark on the horizontal line indicating the severity of the pain they feel. The results will be recorded in mm. Individuals will be asked about their resting activity and nighttime localization and will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Başak KAVALCI KOL, PhD, PT, Principal Investigator — Kirsehir Ahi Evran Universitesi; Merve FIRAT, PhD, PT, Study Chair — Kirsehir Ahi Evran Universitesi; Figen TUNCAY, Prof. Dr., Study Chair — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, 63 / 5.000 Physical Therapy and Rehabilitation Center, Cardiopulmonary Unit, Kırşehir, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data as we store it securely in a locked cabinet and cloud database